CLINICAL TRIAL: NCT06148025
Title: A Human Experimental Medicine Study to Assess Whether the Gut Microbiota Regulates Specific and Non-specific Immune Responses to Vaccination
Brief Title: Antibiotics and Vaccine Immune Responses Study
Acronym: AVIRS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: South Australian Health and Medical Research Institute (Other)
Collaborators: Royal Adelaide Hospital (Other); Flinders University (Other); University of Sydney (Other); Telethon Kids Institute (Other); Centenary Institute (Unknown)
Responsible Party: Principal Investigator, David Lynn, Director, Computational & Systems Biology Program, South Australian Health and Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2023/HREC00066
Record Dates: First submitted 2023-09-29; First posted 2023-11-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-05

CONDITIONS: Vaccine Response Impaired
Keywords: Healthy participants; 18-35 years old; BCG vaccine; Yellow Fever vaccine; Antibiotics
MeSH Terms: interventions — BCG Vaccine; Yellow Fever Vaccine; Vancomycin; Neomycin; Metoclopramide; Loperamide

STUDY DESIGN:
Intervention Model Description: Participants are allocated to Substudy 1 (BCG re-challenge) or Substudy 2 (Yellow Fever vaccine) Participants are randomised to receive
  * antibiotics or comparator (unblinded) and
  * BCG vaccine or placebo (blinded)
  * BCG vaccine or Yellow Fever vaccine (unblinded)
Who Masked: Participant, Investigator
Masking Description: Participants and Investigator are blinded to BCG vaccine or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Substudy 1 - BCG vaccine, antibiotics and 2nd BCG vaccine (Experimental): Randomised to receive antibiotics and a BCG vaccine at visit 1 and a second BCG vaccine 6 months later
  Interventions: Biological: BCG vaccine; Drug: Vancomycin Oral Capsule; Drug: Neomycin Oral Product; Drug: Metoclopramide (Maxolon); Drug: Loperamide HCl
- Substudy 1 - BCG vaccine, no antibiotics and 2nd BCG vaccine (Experimental): Randomised to receive no antibiotics and a BCG vaccine at visit 1 and a second BCG vaccine 6 months later
  Interventions: Biological: BCG vaccine
- Substudy 1 - BCG vaccine, antibiotics and placebo vaccine (Experimental): Randomised to receive antibiotics, a placebo vaccine at visit 1 and a BCG vaccine 6 months later
  Interventions: Biological: BCG vaccine; Drug: Vancomycin Oral Capsule; Drug: Neomycin Oral Product; Drug: Metoclopramide (Maxolon); Drug: Loperamide HCl
- Substudy 1 - BCG vaccine, no antibiotics and placebo vaccine (Experimental): Randomised to receive no antibiotics, a placebo vaccine at visit 1 and a BCG vaccine 6 months later
  Interventions: Biological: BCG vaccine
- Substudy 2 - Yellow Fever vaccine, antibiotics and BCG vaccine (Experimental): Randomised to receive antibiotics, a BCG vaccine at visit 1 and a Yellow Fever vaccine 3 months later
  Interventions: Biological: BCG vaccine; Biological: Yellow Fever vaccine; Drug: Vancomycin Oral Capsule; Drug: Neomycin Oral Product; Drug: Metoclopramide (Maxolon); Drug: Loperamide HCl
- Substudy 2 - Yellow Fever vaccine, no antibiotics and BCG vaccine (Experimental): Randomised to receive no antibiotics, a BCG vaccine at visit 1 and a Yellow Fever vaccine 3 months later
  Interventions: Biological: BCG vaccine; Biological: Yellow Fever vaccine
- Substudy 2 - Yellow Fever vaccine, antibiotics and placebo vaccine (Experimental): Randomised to receive antibiotics, a placebo vaccine at visit 1 and a Yellow Fever vaccine 3 months later
  Interventions: Biological: Yellow Fever vaccine; Drug: Vancomycin Oral Capsule; Drug: Neomycin Oral Product; Drug: Metoclopramide (Maxolon); Drug: Loperamide HCl
- Substudy 2 - Yellow Fever vaccine, no antibiotics and placebo vaccine (Experimental): Randomised to receive no antibiotics, a placebo vaccine at visit 1 and a Yellow Fever vaccine 3 months later
  Interventions: Biological: Yellow Fever vaccine

INTERVENTIONS:
Biological: BCG vaccine — 0.1ml injected intradermally over the distal insertion of the deltoid muscle onto the humerus
  Arms: Substudy 1 - BCG vaccine, antibiotics and 2nd BCG vaccine; Substudy 1 - BCG vaccine, antibiotics and placebo vaccine; Substudy 1 - BCG vaccine, no antibiotics and 2nd BCG vaccine; Substudy 1 - BCG vaccine, no antibiotics and placebo vaccine; Substudy 2 - Yellow Fever vaccine, antibiotics and BCG vaccine; Substudy 2 - Yellow Fever vaccine, no antibiotics and BCG vaccine
Biological: Yellow Fever vaccine — 0.5ml injected subcutaneously
  Arms: Substudy 2 - Yellow Fever vaccine, antibiotics and BCG vaccine; Substudy 2 - Yellow Fever vaccine, antibiotics and placebo vaccine; Substudy 2 - Yellow Fever vaccine, no antibiotics and BCG vaccine; Substudy 2 - Yellow Fever vaccine, no antibiotics and placebo vaccine
Drug: Vancomycin Oral Capsule — 500mg every 6 hours for 3 days
  Other Names: Firvanq; Vancocin HCl Pulvules
  Arms: Substudy 1 - BCG vaccine, antibiotics and 2nd BCG vaccine; Substudy 1 - BCG vaccine, antibiotics and placebo vaccine; Substudy 2 - Yellow Fever vaccine, antibiotics and BCG vaccine; Substudy 2 - Yellow Fever vaccine, antibiotics and placebo vaccine
Drug: Neomycin Oral Product — 1000mg every 6 hours for 3 days
  Other Names: Neo-Fradin
  Arms: Substudy 1 - BCG vaccine, antibiotics and 2nd BCG vaccine; Substudy 1 - BCG vaccine, antibiotics and placebo vaccine; Substudy 2 - Yellow Fever vaccine, antibiotics and BCG vaccine; Substudy 2 - Yellow Fever vaccine, antibiotics and placebo vaccine
Drug: Metoclopramide (Maxolon) — 10mg every 8 hours
  Arms: Substudy 1 - BCG vaccine, antibiotics and 2nd BCG vaccine; Substudy 1 - BCG vaccine, antibiotics and placebo vaccine; Substudy 2 - Yellow Fever vaccine, antibiotics and BCG vaccine; Substudy 2 - Yellow Fever vaccine, antibiotics and placebo vaccine
Drug: Loperamide HCl — 2mg tablets/capsules: 2 tablets/capsules initially, followed by 1 tablet after each loose motion, to a maximum of 8 tablets/capsules per day
  Arms: Substudy 1 - BCG vaccine, antibiotics and 2nd BCG vaccine; Substudy 1 - BCG vaccine, antibiotics and placebo vaccine; Substudy 2 - Yellow Fever vaccine, antibiotics and BCG vaccine; Substudy 2 - Yellow Fever vaccine, antibiotics and placebo vaccine

SUMMARY:
The goal of this clinical trial is to examine immune responses to the BCG vaccine in healthy adults who have, or who have not, taken antibiotics to deplete their gut bacteria prior to vaccination.

The main question it aims to answer is: does depletion of the gut microbiota lead to impaired BCG-induced protection against specific and non-specific to challenges to the immune system?

DETAILED DESCRIPTION:
The study is divided into two sub-studies. The first sub-study (BCG re-challenge) is an experimental medicine study in 168 healthy participants to determine if depletion of the gut microbiota leads to impaired BCG-induced protection against a subsequent Mycobacterium bovis BCG intradermal challenge.

The second sub-study (Yellow Fever vaccine) has a very similar experimental design to the first but will determine if depletion of the gut microbiota leads to impaired BCG-induced protection against other infections. To assess this, participants in this sub-study (n=180) will be re-challenged after 3 months with a live attenuated viral vaccine, the Yellow Fever vaccine, which induces a mild viremia.

In both sub-studies, participants will initially be randomised to receive a 3 day course of antibiotics or none (comparator group). The two groups in each sub-study will be randomised again to receive either BCG vaccine or 0.9% NaCl placebo injection in the left arm.

BCG re-challenge sub-study (Sub-study 1): Six months following randomisation, all participants will receive a BCG vaccine challenge in the right arm. A punch skin biopsy will be taken of this challenge site 2 weeks after the challenge to assess M. bovis BCG bacterial load in the skin.

Yellow Fever vaccine sub-study (Sub-study 2): Three months following randomisation, all participants will receive a Yellow Fever vaccine challenge in the right arm. Blood samples will be collected from Yellow Fever vaccinated participants at day 3, 5 and 7 following Yellow Fever vaccine challenge to quantify Yellow Fever viral load in blood.

All participants in both sub-studies will have blood samples collected at randomisation, before each vaccination, 2 weeks after each BCG vaccination and in the Yellow Fever vaccine sub-study at day 3, 5 and 7 following Yellow Fever vaccination. Stool samples will be collected prior to randomisation, and prior to each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Provided a signed and dated informed consent form
* BCG naïve (Arm 1) and BCG and YF vaccine naïve (Arm 2)
* Willing to take short antibiotic course
* Willing to undergo a punch biopsy (Arm 1)
* Willing to have up to 7 blood samples and 3 stool samples collected over 5-7 months
* Not pregnant or intending to get pregnant for the duration of the study (a pregnancy test will be offered to females)

Exclusion Criteria:

* Previous BCG or YF vaccination
* Previous YF infection
* Evidence of latent TB infection (LTBI) (assessed through a questionnaire) (IGRA to confirm if needed)
* People with contraindications for BCG vaccination:

  * malignancies involving bone marrow or lymphoid systems, primary or secondary immunodeficiencies, HIV infection
  * moderate/severe skin disease including eczema, dermatitis or psoriasis
  * requiring immunosuppressive drugs or other immune modifying drugs e.g. corticosteroids, non-biological immunosuppressants, biological agents (such as monoclonal antibodies against tumour necrosis factor (TNF)-alpha)
* People with contraindications to YF vaccination:

  * History of thymus disease, including myasthenia gravis, thymoma, thymectomy, DiGeorge syndrome, thymic damage from chemoradiotherapy or graft-versus-host disease
  * YF vaccination is contraindicated in immunocompromised individuals, including individuals who have HIV infection, primary immunodeficiencies (including inherited IFNAR1 deficiency), or are taking corticosteroids or other immunosuppressive agents and haematopoietic stem cell transplant recipients
  * People who have had a haematopoietic stem cell transplant
  * Individuals with history of severe allergic reactions to egg or chicken proteins
* Pregnant or breastfeeding or planning to become pregnant
* History of renal disease/insufficiency
* Tattoo obscuring BCG vaccination site(s)
* Any history of severe allergic reaction or anaphylaxis to vaccination or antibiotics
* People with chronic serious underlying illness
* Have received any prescribed oral or intravenous antibiotic in the 28 days prior to study visits 1 and 4 (including isoniazid, rifampicin, streptomycin and ethambutol as these particular antibiotics have activity against M. bovis)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 348 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Sub-study 1 BCG re-challenge | 5 years
  Mycobacterial load (Colony Forming Units (CFU)) in the skin biopsy site in BCG-vaccinated participants not exposed to antibiotics (BCG-No ABX) compared to BCG-vaccinated participants that were exposed to antibiotics (BCG-ABX)
Sub-study 2 Yellow Fever vaccine | 5 years
  Yellow Fever viremia (viral copies/ml blood) at D3-7 post YF vaccination in BCG-vaccinated participants not exposed to antibiotics (BCG-No ABX) compared to BCG-vaccinated participants that were exposed to antibiotics (BCG-ABX)

SECONDARY OUTCOMES:
Sub-study 1 - Bacterial load | 5 years
  Day 0 bacterial load (16S copies/g stool) in all ABX participants vs No-ABX participants
Sub-study 2 - Bacterial load | 5 years
  Day 0 bacterial load (16S copies/g stool) in all ABX participants vs No-ABX participants
Sub-study 1 - Microbiota diversity | 5 years
  Day 0 microbiota diversity (Shannon diversity index) in all ABX participants vs No-ABX participants
Sub-study 2 - Microbiota diversity | 5 years
  Day 0 microbiota diversity (Shannon diversity index) in all ABX participants vs No-ABX participants
Sub-study 1 - Mycobacterial load | 5 years
  Mycobacterial load (CFU) in the skin biopsy site in BCG-vaccinated participants compared to placebo-vaccinated participants
Sub-study 1 - Mycobacterial IFNγ responses | 5 years
  IFNγ production in pg/mL following stimulation of PBMC with mycobacteria in BCG-ABX participants versus BCG-No ABX participants
Sub-study 1 - Mycobacterial T cell activation marker responses | 5 years
  % of CD69+CD137+ CD4 T cells following stimulation of PBMC with mycobacteria in BCG-ABX participants versus BCG-No ABX participants
Sub-study 2 - Peak viraemia | 5 years
  Peak viraemia (viral copies/ml blood) at D3-7 post YF vaccination in BCG-vaccinated participants compared to placebo-vaccinated participants
Sub-study 2 - Heterologous TNFα responses following R848 stimulation | 5 years
  D90 PBMC TNFα responses (pg/mL) following in vitro stimulation with viral ligand R848 in BCG-ABX participants versus BCG-No ABX participants
Sub-study 2 - Heterologous TNFα responses following LPS stimulation | 5 years
  D90 PBMC TNFα responses (pg/mL) following in vitro stimulation with bacterial ligand LPS in BCG-ABX participants versus BCG-No ABX participants
Sub-study 2 - Heterologous TNFα responses following fungal stimulation | 5 years
  D90 PBMC TNFα responses (pg/mL) following in vitro stimulation with fungal ligand heat-killed C. albicans in BCG-ABX participants versus BCG-No ABX participant

CONTACTS AND LOCATIONS:
Overall Officials: Simone Barry, Principal Investigator — Royal Adelaide Hospital; David Lynn, Principal Investigator — South Australian Health and Medical Research Institute
Locations (1):
- South Australian Health and Medical Research Institute, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable individual participant data from the study may be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept SAHMRI's conditions, under a collaborator agreement, for accessing:
  * Individual participant data that underlie the results reported in our articles after deidentification (text, tables, figures and appendices)
  * Study protocol, Statistical Analysis Plan, PICF
  Molecular data generated from this study (i.e. transcriptomic, epigenomic and metagenomic) will be labelled with a unique identification code and stored on an appropriate data repository (e.g. Gene Expression Omnibus, Sequence Read Archive) with demographic information (age and sex). No identifying participant information will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At time of publication. Data will be available indefinitely.
Access Criteria: Researchers from a recognised research institution can approach SAHMRI for access of data. The researcher will need to provide evidence that the proposed use of the data has been ethically reviewed and approved by an Institutional Review Board (IRB)/ Human Research Ethics Committee(HREC), and accept SAHMRI's conditions, under a collaborator agreement.